CLINICAL TRIAL: NCT04878471
Title: A Phase 1 Single Intravenous Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ASP5354 in Healthy Adult Japanese Male Participants
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ASP5354 in Healthy Adult Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 5354-CL-0002; jRCT2071210026 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-05-06; First posted 2021-05-07 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
Keywords: ASP5354; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASP5354 (Experimental): Three participants in three dose levels will receive a single intravenous dose of ASP5354 on Day 1 under fasting conditions.
  Interventions: Drug: Pudexacianinium chloride
- ASP5354 Matching Placebo (Placebo Comparator): One participant in three dose levels will receive a single intravenous dose of matching placebo on Day 1 under fasting conditions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pudexacianinium chloride — Intravenous
  Other Names: ASP5354
  Arms: ASP5354
Drug: Placebo — Intravenous
  Arms: ASP5354 Matching Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of single intravenous doses of ASP5354 in healthy, adult Japanese male participants.

DETAILED DESCRIPTION:
This study is comprised of 3 parts. Part 1 and Part 2 will be conducted in a parallel manner while Part 3 will be conducted subsequentially. Participants will be residential for a period of 3 days/2 nights. Participants will be discharged from the clinical unit on day 2 on the condition that all required assessments have been performed and that there are no medical reasons for a longer stay in the clinical unit.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index (BMI) range of 17.6 to 26.4 kg/m^2 inclusive and weighs at least 50 kg at screening.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 30 days after Investigational Product (IP) administration.
* Male participant must not donate sperm during the treatment period and for 30 days after IP administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after IP administration.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has received any investigational therapy within 12 weeks prior to screening.
* Participant has any condition that makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP5354 or any components of the formulation used.
* Participant has had previous exposure with ASP5354.
* Participant has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST] and total bilirubin [TBL]) above the upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Participant has creatinine level outside normal limits on day -1. In such a case, the assessment may be repeated once.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to IP administration.
* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Participant has any clinically significant abnormality following the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or on day -1.
* Participant has a mean pulse < 40 or > 100 bpm; mean systolic blood pressure (SBP) < 90 or > 140 mmHg; mean diastolic blood pressure (DBP) < 40 or > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day-1. If the mean blood pressure exceeds the limits above, one additional triplicate may be taken.
* Participant has body temperature < 35.0ºC or >= 37.5ºC on day -1.
* Participant has a mean corrected QT interval using Fridericia's formula (QTcF) of > 430 msec on day -1. If the mean QTcF exceeds the limits above, one additional triplicate ECG may be taken.
* Participant has used any prescribed or nonprescribed drugs (including vitamins, oral contraceptives or hormone replacement therapy (HRT) and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to IP administration, except for occasional use of acetaminophen (up to 2 g/day) and topical dermatological products (including corticosteroid products).
* Participant has a history of smoking > 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to day -1.
* Participant has a history of consuming > 16 units of alcohol per week within 3 months prior to day -1 (note: 1 unit = 10 g pure alcohol, = 250 mL of beer [5%], 35 mL of spirits [35%] or 100 mL of wine [12%]).
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or morphine and phencyclidines) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and morphine, phencyclidines) at screening or on day -1.
* Participant has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Participant has had significant blood loss, donated >= 400 mL of whole blood within 90 days, >= 200 mL of whole blood within 30 days or donated blood components within 14 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Participant has a positive serology test for hepatitis B core (HBc) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies and antigen or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 and syphilis at screening.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 6 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study investigational product (IP), whether or not considered related to the study IP. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or requires medical or surgical intervention to prevent one of the other outcomes listed above.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 6 days
  Number of participants with potentially clinically significant laboratory values
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to 6 days
  Number of participants with potentially clinically significant vital sign values
Number of participants with routine 12-lead electrocardiogram (ECG) abnormalities and/or adverse events (AEs) | Up to 6 days
  Number of participants with potentially clinically significant ECG values

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP5354 in plasma: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Up to 2 days
  AUCinf will be recorded from the pharmacokinetic (PK) plasma samples collected
PK of ASP5354 in plasma: Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Up to 2 days
  AUClast will be recorded from the PK plasma samples collected
PK of ASP5354 in plasma: Maximum concentration (Cmax) | Up to 2 days
  Cmax will be recorded from the PK plasma samples collected
PK of ASP5354 in urine: amount of administered dose excreted from the time of dosing to the last measurable point after dosing | Up to 2 days
  Aelast will be recorded from the PK urine samples collected
PK of ASP5354 in urine: percent of administered dose excreted from the time of dosing to the last measurable point after dosing | Up to 2 days
  Aelast% will be recorded from the PK urine samples collected
PK of ASP5354 in urine: Renal Clearance (CLR) | Up to 2 days
  CLR will be recorded from the PK urine samples collected

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- JP81001, Sumida-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.